CLINICAL TRIAL: NCT04772885
Title: A Phase 1 Randomized, Placebo-controlled, Single and Multiple Ascending Dose Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Orally Administered KT-474 in Healthy Adult Volunteers and Patients With Atopic Dermatitis (AD) or Hidradenitis Suppurativa (HS)
Brief Title: A Single and Multiple Ascending Dose Trial of KT-474 in Healthy Adult Volunteers and Patients With Atopic Dermatitis (AD) or Hidradenitis Suppurativa (HS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kymera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KT474-HV-101
Record Dates: First submitted 2021-02-12; First posted 2021-02-26 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteer; Atopic Dermatitis; Hidradenitis Suppurativa
Keywords: Atopic Dermatitis; Hidradenitis Suppurativa; Immune-inflammatory diseases
MeSH Terms: conditions — Dermatitis, Atopic; Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: Single ascending dose escalation and multiple ascending dose escalation study followed by an evaluation of food effects on absorption
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomized double blind (for Parts A and B only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single ascending dose cohorts in healthy subjects (Experimental): Healthy volunteer subject cohorts randomized 6:2 receiving a single dose of KT-474 or placebo. The first cohort will receive 25 mg of KT-474 or placebo. Dose escalation will occur if KT-474 or placebo is tolerated.
  Interventions: Drug: KT-474/Placebo
- Multiple ascending dose cohorts in healthy subjects (Experimental): Healthy volunteer subject cohorts randomized 9:3 to receive KT-474 or placebo for 14 days continuous dosing. The first cohort will receive a dose of KT-474 or placebo determined to be safe based on data generated in the SAD portion.
  Interventions: Drug: KT-474/Placebo
- Food Effect Cohort in healthy subjects (Experimental): Healthy Volunteer SAD subject cohorts (up to 5) will receive a single dose of KT-474 in the fed state.
  Interventions: Drug: KT-474/Placebo
- Multiple dose cohort in HS and AD patients (Experimental): A single cohort of up to 30 patients with AD or HS to receive a dose of KT-474 determined to be safe based on data generated in the healthy volunteer MAD portion, dosed daily X 28 days.
  Interventions: Drug: KT-474
- Multiple dose cohorts in healthy subjects (Experimental): Healthy volunteer subject cohorts randomized 9:3 to receive KT-474 or placebo every other day over 14 days, and/or twice weekly over 15 days. The first cohort will receive a dose of KT-474 or placebo determined to be safe based on data generated in the SAD and MAD portion.
  Interventions: Drug: KT-474/Placebo

INTERVENTIONS:
Drug: KT-474/Placebo — KT-474 or matching placebo oral tablet(s)
  Arms: Food Effect Cohort in healthy subjects; Multiple ascending dose cohorts in healthy subjects; Multiple dose cohorts in healthy subjects; Single ascending dose cohorts in healthy subjects
Drug: KT-474 — KT-474 oral tablet(s)
  Arms: Multiple dose cohort in HS and AD patients

SUMMARY:
KT-474 is an oral heterobifunctional small molecule IRAK4 degrader being developed for the treatment of interleukin-1 receptor (IL-1R)/toll-like receptor (TLR)-driven immune-inflammatory diseases. This first-in-human (FIH) study will characterize the safety, tolerability and the pharmacokinetics/pharmacodynamics (PK/PD) of a single ascending dose and multiple ascending doses of KT-474 in healthy volunteers and patients with atopic dermatitis (AD) or hidradenitis suppurativa (HS). The effects of food on the absorption of KT-474 will also be evaluated in healthy volunteers.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1 randomized, placebo-controlled, single and multiple ascending dose trial of KT-474 that will characterize the safety, PK and PD of orally administered KT-474 after a single dose (Part A) and after repeated dosing first in healthy adult volunteers (Part B) and then in patients with AD or HS (Part C). Initially, a dose range of KT-474 in single ascending dose (SAD) escalation cohorts will be explored in healthy subjects. Up to five single dose cohorts of healthy subjects is also planned to understand food effects (FE) on the PK of KT-474. Enrollment of healthy subjects into 2-week multiple ascending dose (MAD) escalation cohorts will be initiated once sufficient safety and PK data from multiple SAD cohorts are available to inform the safe starting dose for the 2-week MAD portion of the study. After the MAD portion in healthy subjects is completed, the safety, PK, and PD of a dose of KT-474 that was found to be safe in healthy subjects when administered for 2 weeks will then be evaluated in AD or HS subjects for 28 days of dosing. Separately, additional multiple dose cohorts evaluating once every other day and/or twice weekly dosing schedules at or below previously evaluated dose levels in healthy volunteers may be initiated.

ELIGIBILITY:
Healthy Volunteer (Parts A and B) Inclusion Criteria:

1. Male and female subjects, including female subjects of child bearing potential, between the ages of 18 and 55 with a weight at least 50 kg and a body mass index (BMI) between 18.0 and 30.0 kg/m2.
2. Subjects confirmed as negative in severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection test at Screening and on Day -2.
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Agreement and ability to comply with all contraception requirements if applicable.
5. All subjects must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Healthy Volunteer (Parts A and B) Exclusion Criteria:

1. Evidence or history of a clinically significant medical condition or other condition that might significantly interfere with the absorption, distribution, metabolism, or excretion of study drug, or place the subject at an unacceptable risk as a participant in this study.
2. Healthy volunteers who have a clinically relevant history or presence of respiratory, GI, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, or connective tissue diseases or disorders.
3. Healthy volunteers who have any known factor, condition, or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease.
4. Female Healthy volunteers who are pregnant, trying to become pregnant or lactating or breastfeeding.
5. Healthy volunteers who have participated in any investigational drug or device clinical study within 3 months prior to first dosing on this study.
6. Healthy volunteers who have previously participated in a study with an investigational product or device involving the dosing of a biological targeted at any immune pathway within 1 year prior to Screening.

AD or HS Patient (Part C) Inclusion Criteria:

1. Male or female patients aged 18 years to 55 years (inclusive) at the time of Screening, and in generally good health, except for AD or HS, and has a BMI of 17.5 to 35.0 kg/m2; and a total body weight >50 kg (110 lb).
2. Diagnosis of AD or HS for at least 6 months.
3. Patients with AD: having at least 10% treatable percentage body surface area at Screening or on Admission (excluding the scalp and designated venous access areas).
4. Willingness and ability to comply with all contraception requirements as applicable based on reproductive status.
5. Has adequate venous access with venous access sites having AD-unaffected, non-infected skin to permit repeated PK sampling.
6. Female patients must have a negative result for the serum pregnancy test at the Screening Visit and on admission.
7. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
8. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
9. Patients with HS: A total Abscess and Inflammatory Nodule count of ≥4 at baseline

AD or HS Patient (Parts C) Exclusion Criteria:

1. Has any clinically significant medical disorder, condition, disease (including active or potentially recurrent dermatological conditions other than AD or HS), significant physical examination or laboratory findings that may interfere with study objectives, in the Investigator's opinion (eg, conditions or findings that may expose a patient to unacceptable risk by study participation, confound the evaluation of treatment response or adverse events, or otherwise interfere with a patient's ability to complete the study).
2. Has an active systemic or soft tissue infection, including known actively-infected AD or HS skin lesion.
3. Treatment with an investigational product within 30 days or 5 half-lives preceding the first dose of investigational product (whichever is longer).
4. Use of prescription or nonprescription drugs including topical corticosteroids, vitaminic and dietary supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
5. Blood donation (excluding plasma donations and platelet donations) of approximately ≥400 mL within 3 months or ≥200 mL within a month prior to dosing.
6. History of sensitivity to heparin or heparin-induced thrombocytopenia.
7. Unwilling or unable to comply with the protocol procedures and/or assessments.
8. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for entry into this study.
9. Patients with HS: Fistula and Tunnel count of >20 at baseline.
10. Patients with AD: Active herpes infection or history of eczema herpeticum.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent Adverse Events | up to 28 days
Incidence and frequency of use of concomitant medication | up to 28 days

SECONDARY OUTCOMES:
Area under the curve plasma concentration from time zero to infinity [AUC(0-∞)] (single dose only) | up to 28 days
Area under the curve plasma concentration from time zero to last measurable concentration [AUC(0-last)] | up to 28 days
Area under the plasma concentration-time curve during a dosing interval [AUC(0-tau)] | up to 28 days
Maximum observed plasma concentration (Cmax) | up to 28 days
Time to maximum observed plasma concentration (Tmax) | up to 28 days
Apparent clearance (CL/F) | up to 28 days
Apparent volume of distribution (Vz/F) | up to 28 days
Terminal elimination half-life (t1/2) | up to 28 days
Mean residence time (MRT) | up to 28 days
Renal clearance (CLR) | up to 28 days

OTHER OUTCOMES:
IRAK4 levels in peripheral blood mononuclear cells | up to 28 days
IRAK4 levels in skin | up to 28 days
Percentage Change from baseline in Total Abscess and Inflammatory Nodule (AN) Count, Skin Pain Numerical Rating Scale (NRS), Peak pruritis NRS, and HS Physician's Global Assessment (HS-PGA) in HS patients | up to 42 days
Percentage Change from baseline in Eczema Area and Severity Index (EASI), Peak Pruritus Numerical Rating Scale (NRS) and Investigator Global Assessment (IGA) in AD patients | up to 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Gollerkeri, MD, Study Director — Kymera Therapeutics, Inc.
Locations (14):
- United States (14):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Southwest Skin Specialists 32nd St, Phoenix, Arizona
  - Southwest Skin Specialists Tatum, Phoenix, Arizona
  - Beatrice Keller Clinic, Sun City West, Arizona
  - Encore Medical Research, LLC. - Boynton Beach, Boynton Beach, Florida
  - Research Centers of America, Hollywood, Florida
  - Encore Medical Research, LLC. - Hollywood, Hollywood, Florida
  - Encore Medical Research, LLC. - Weston, Weston, Florida
  - Dermatology and Skin Cancer Center of Leawood, Leawood, Kansas
  - Dermatology and Skin Cancer Center of Overland Park, Overland Park, Kansas
  - Dermatology and Skin Cancer Center of Lee's Summit, Lee's Summit, Missouri
  - TKL Research, Fair Lawn, New Jersey
  - U.S. Dermatology Partners Jollyville, Austin, Texas
  - U.S. Dermatology Partners Cedar Park, Cedar Park, Texas

REFERENCES:
- [Derived] Ackerman L, Acloque G, Bacchelli S, Schwartz H, Feinstein BJ, La Stella P, Alavi A, Gollerkeri A, Davis J, Campbell V, McDonald A, Agarwal S, Karnik R, Shi K, Mishkin A, Culbertson J, Klaus C, Enerson B, Massa V, Kuhn E, Sharma K, Keaney E, Barnes R, Chen D, Zheng X, Rong H, Sabesan V, Ho C, Mainolfi N, Slavin A, Gollob JA. IRAK4 degrader in hidradenitis suppurativa and atopic dermatitis: a phase 1 trial. Nat Med. 2023 Dec;29(12):3127-3136. doi: 10.1038/s41591-023-02635-7. Epub 2023 Nov 13. PMID 37957373